CLINICAL TRIAL: NCT01899573
Title: A Study of Percutaneous Left Ventricular Reshaping of Mitral Apparatus to Reduce Functional Mitral Regurgitation and Improve LV Function Using the Accucinch® System
Brief Title: Percutaneous Left Ventricular Reshaping to Reduce Functional Mitral Regurgitation and Improve LV Function
Acronym: LVRESTORESA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ancora Heart, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3566
Record Dates: First submitted 2013-07-03; First posted 2013-07-15 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Functional Mitral Regurgitation
Keywords: Heart failure; mitral regurgitation; mitral valve
MeSH Terms: conditions — Heart Failure; Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Device: AccuCinch® Ventriculoplasty System

INTERVENTIONS:
Device: AccuCinch® Ventriculoplasty System — Percutaneous intervention for the treatment of functional mitral regurgitation

SUMMARY:
The study is designed to demonstrate the safety, feasibility and potential efficacy of using the AccuCinch® System to reduce functional mitral regurgitation.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Subjects with clinically significant mitral regurgitation (MR 2+ and above)
* Ejection Fraction ≥ 25%
* Stable cardiac medical regimen for heart failure for at least 1 month
* Stable NYHA Classification for at least 1 month
* Subject is eligible for cardiac surgery
* The subject has been informed of the nature of the study, agrees to its provisions, and has provided written informed consent

Exclusion Criteria:

* Myocardial infarction within 90 days of the intended treatment with the device
* Prior surgical, transcatheter, or percutaneous mitral valve intervention
* Any intervention for coronary artery disease (CAD) within the last 30 days prior to treatment, or unrevascularized multivessel coronary disease
* Hemodynamic instability or the need for emergent surgery
* Non-ambulatory NYHA Class IV symptoms of heart failure or subjects requiring IV inotropic support
* Subjects in whom sufficient quality of echocardiography (TTE and TEE) cannot be obtained
* Echocardiography evidence of primary mitral valve disease causing MR or MS,
* Evidence of mitral valve stenosis with an estimated valve area less than 3.0 cm2
* Mitral valve prosthesis or pathology that would prevent adequate function of the GDS Accucinch System
* Estimated GFR of <30ml/min/1.73m2
* Greater than mild mitral annular calcification observed by fluoroscopy
* Presence of aortic valve prosthesis
* Moderate to severe aortic valve stenosis or calcification observed by echocardiography or fluoroscopy
* Severe aortic arch calcification or mobile aortic atheroma observed by echocardiography or fluoroscopy
* Active bacterial endocarditis
* History of bleeding diathesis or coagulopathy
* History of stroke within the prior 6 months
* Subjects in whom anticoagulation is contraindicated
* Any clinical evidence that the investigator feels would place the subject at increased risk with the placement of the device.
* Concurrent medical condition with a life expectancy of less than 12 months
* Currently participating in an investigational study
* Co-morbid conditions that place the subject at an unacceptable surgical risk (e.g. severe chronic obstructive pulmonary disease, hepatic failure, immunological abnormalities, and hematological abnormalities)
* Subjects with indication for concomitant surgery such as coronary artery bypass graft (CABG), aortic valve reconstruction or replacement, tricuspid repair or replacement, left ventricular remodeling surgery and congenital repair
* Any cardiac resynchronization therapy within the last 3 months prior to treatment
* Subjects on high dose steroids or immunosuppressant therapy
* Female subjects who are pregnant, of child bearing potential or lactating
* Subjects who are unable or unwilling to comply with the follow-up schedule and requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-10; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac and cardiovascular events | 30 day

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica CardioVID, Medellín, Colombia